CLINICAL TRIAL: NCT01062815
Title: Prevention of Parenteral Nutrition-Associated Cholestasis With Cyclic Parenteral Nutrition in Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Lesley Smith, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20080651
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Cholestasis; Prematurity; Gastroschisis; Intestinal Atresia; Necrotizing Enterocolitis
Keywords: PNALD; PNAC; Parenteral Nutrition-Associated Cholestasis; Congenital Anomalies of Gastrointestinal Tract
MeSH Terms: conditions — Cholestasis; Premature Birth; Gastroschisis; Intestinal Atresia; Enterocolitis, Necrotizing | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycling Parenteral Nutrition (Experimental): Infants in the intervention cycling group will receive infusion of carbohydrate/amino acids and intralipid over a 20-hour period. During the 4-hour window period, infants in this group will receive dextrose solution only at the same rate calculated for the carbohydrate/amino acid infusion.
  Interventions: Dietary Supplement: Parenteral Nutrition
- Continuous Parenteral Nutrition (Active Comparator): Infants in this control group will receive infusion of carbohydrates/amino acids and intralipids continuously, over 24 hours.
  Interventions: Dietary Supplement: Parenteral Nutrition

INTERVENTIONS:
Dietary Supplement: Parenteral Nutrition — Parenteral Nutrition infused over 20 hours cycled with dextrose solution over 4 hours compared to Parenteral Nutrition infused continuously over 24 hours.

SUMMARY:
Hypothesis to be Tested:

Since the first description of intravenous alimentation over half a century ago, parenteral nutrition (PN) has become a common nutritional intervention for conditions characterized by inability to tolerate enteral feeds such as Short Bowel Syndrome, Chronic Intestinal Pseudoobstruction, Microvillus Inclusion Disease, Crohn's disease, multi-organ failure and prematurity. Parenteral Nutrition-Associated Liver Disease (PNALD) encompasses a spectrum of disease including cholestasis, hepatitis, steatosis and gallbladder sludge/stones which may progress to liver cirrhosis and even failure.

There is a direct correlation between duration of parenteral nutrition and development of cholestasis in infants. There is evidence in animals and humans that cycling of parental nutrition, defined as infusing nutrients over a time period shorter than 24 hours, reduces cholestasis. There is also data that premature infants with gestational age (GA) < 32 weeks and birth weight <1500g, as well as infants with congenital anomalies of the gastrointestinal tract, are among those at highest risk of developing Parenteral Nutrition-Associated Cholestasis (PNAC).

We therefore hypothesize that infants with gestational age (GA) <32 weeks and birth weight (BW) between <1500g, or with congenital anomaly of the gastrointestinal tract regardless of GA or BW, receiving PN over a period of 20 hours will have a decrease severity of PNAC, demonstrated by a lower peak direct bilirubin, compared to a similar control population receiving standard 24 hour infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Infants expected to need prolonged PN (receiving >75% PN on dol 7) with the following risk factors:

   1. Prematurity with gestational age (GA) <32 weeks AND birth weight <1500g. OR
   2. Congenital anomaly of the gastrointestinal tract regardless of GA or BW
2. Screening direct bilirubin prior to the initiation of parenteral nutrition <2mg/dL.

Exclusion Criteria:

1. Infants with major congenital anomalies, other than those of the gastrointestinal tract.
2. Infants with known obstruction of the hepatobiliary tract.
3. Infants with suspected congenital infection or suspected genetic/metabolic syndrome predisposing them to cholestasis based on direct bilirubin > 2mg/dL prior to instituting PN.

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a decreased peak direct bilirubin in infants with GA <32 weeks and BW between <1500g, or with congenital anomaly of the gastrointestinal tract regardless of GA or BW, requiring prolonged PN (receiving >75% PN on dol 7). | Peak direct bilirubin during time period: Initiation to Discontinuation of PN (Defined as successfully off PN for 7days)

SECONDARY OUTCOMES:
A secondary outcome is to determine if the incidence of PN- Associated Cholestasis is lower in infants receiving cyclic PN over 20 hours compared to infants receiving standard continuous PN over 24 hours. | Incidence of cholestasis (direct bilirubin >2mg/dL) during time period: Initiation to Discontinuation of PN (Defined as successfully off PN for 7days)
A secondary outcome in infants who develop PN-Associated Cholestasis is to evaluate if those receiving cyclic PN will have a shorter duration of cholestasis compared to infants receiving continuous PN. | Duration of cholestasis (# of days direct bilirubin > 2mg/dL) during time period: Initiation to Discontinuation of PN (Defined as successfully off PN for 7days) .
A secondary outcome is to evaluate if infants receiving cyclic PN will have equivalent rates of growth compared to infants receiving continuous PN. | Rate of growth (g of weight and cm of length and head circumference gained per week) during time period: Initiation to Discontinuation of PN (Defined as successfully off PN for 7days).

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Smith, MD, MBA, Principal Investigator — University of Miami, Dept of Pediatrics, Division of GI, Hepatology and Nutrition; Jennifer Garcia, MD, Study Director — University of Miami, Dept of Pediatrics, Division of GI, Hepatology and Nutrition; Teresa DelMoral, MD MPH, Study Chair — University of Miami, Dept of Pediatrics, Division of Neonatology
Locations (1):
- Holtz's Children's Hospital- University of Miami/Jackson Memorial Hospital, Miami, Florida, United States

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765